CLINICAL TRIAL: NCT03841136
Title: Phase II Clinical Trial of Anlotinib Combined With Etoposide and Platinum in the Treatment of Extensive Stage Small Cell Lung Cancer
Brief Title: Anlotinib Combined With Etoposide and Platinum in the Treatment of Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Attending, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-SCLC-001
Record Dates: First submitted 2019-02-01; First posted 2019-02-15 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; Etoposide; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib combined with EP (Experimental): anlotinib combined with etoposide and platinum
  Interventions: Drug: anlotinib

INTERVENTIONS:
Drug: anlotinib — anlotinib 12mg PO QD CBP(AUC 5mg/mL/min，or DDP（75mg/m2）D1 etoposide（100mg/m2）D1~D3
  Other Names: etoposide and platinum

SUMMARY:
To evaluate the progression free survival of patients with extensive stage small cell lung cancer treated with anlotinib combined with EP/CE regimen

DETAILED DESCRIPTION:
To evaluate the progression free survival of patients with extensive stage small cell lung cancer treated with anlotinib combined with EP/CE regimen To evaluate the safety, tolerability, overall survival (OS), objective response rate (ORR), disease control rate (DCR), and quality of life (QoL) of patients with extensive stage small cell lung cancer treated with anlotinib

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in the study and have signed the informed consent.
2. Histological or cytological diagnosis of extensive small cell lung cancer, and no indication of radical surgery or radiotherapy.
3. There are measurable lesions defined by RECIST standard v1.1. A lesion can be considered measurable only if the previously irradiated lesion has clear progression after radiotherapy and the previous irradiated lesion is not the sole lesion.
4. Initially treated patients who have not received any systematic therapy before. If have received postoperative adjuvant chemotherapy, the time to relapse is at least 6 months from the last adjuvant chemotherapy.

5）18~75 years old; ECOG PS score: 0~1 points; expected survival time is more than 3 months.

6）The main organs's function meets the following criteria within 14 days before treatment:

1. Routine blood test (without blood transfusion within 14 days): a) Hemoglobin (HB) ≥ 90 g / L; b) Absolute neutrophil (ANC) ≥ 1.5 × 109 / L; c) Platelets (PLT) ≥ 80×109/L
2. Biochemical examination: a) Total bilirubin (TBIL) ≤ 1.5 times of the upper limit of the normal (ULN); b) Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5ULN.To patients with liver metastasis, ALT and AST ≤ 5ULN; c) Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min;
3. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ the lower limit of the normal (50%).

7）Patients with previously treated asymptomatic CNS metastases are allowed to participate in this study if all of the following criteria are met: a) No need for continuous corticosteroid therapy for CNS disease; b) No radiotherapy within 7 days prior to enrollment treatment; c) Imaging examination from the end of radiotherapy to screening period shows no CNS progression.

8）Women of childbearing age should agree to conduct contraception (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the end of the study; and the serum or urine pregnancy test is negative within 7 days prior to study enrollment and they must be non-lactating patients; Men should agree to conduct contraception during the study and within 6 months after the end of the study.

Exclusion Criteria:

1. Patients who have been treated with anlotinib capsules in the past.
2. Patients who have previously received systemic chemotherapy, signal transduction inhibitors, targeted therapies, hormone and endocrine therapy.
3. Patients with other malignant tumors occurred within 5 years prior to the enrollment, except those with cured cervical carcinoma in situ and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)] , basal or squamous cell skin cancer, and localized prostate cancer and ductal breast carcinoma in situ treated with radical surgery.
4. Unresolved toxicity due to any previous treatment above CTC AE (4.0) level 2 or higher, excluding hair loss.
5. Patients with a variety of factors affecting oral medications (such as dyspahgia, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.)
6. Patients with symptomatic CNS metastases.
7. Patients with dysfucitonal coagulation (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), and bleeding tendency (the following condition must be met within 14 days before the enrollment: the INR is within the normal range without using anticoagulants); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or the like; Patients with International Normalized Ratio (INR) of less than1.5 are allowed to use low-dose warfarin (1 mg orally, once daily) or aspirin (with a daily dose of no more than 100 mg) for prophylactic purposes.
8. Patients with major surgical treatment, incisional biopsy or tremendous traumatic injury within 28 days prior to the enrollment.
9. Patients with tumors that have invaded tissues surrounding vital blood vessels founded in imaging or with a high probability of fatal bleeding due to the invasion of tumors to vital blood vessels according to the judgements of the researchers during the follow-up study.
10. Patients with uncontrolled pleural, pericardial, or peritoneal effusion requiring repeated drainage.
11. Patients with any severe and/or uncontrolled disease, including:

    1. Patients with unsatisfactory blood pressure control (systolic blood pressure >150 mmHg, diastolic blood pressure >90 mmHg).
    2. Patients with myocardial ischemia or myocardial infarction of Grade I of higher level, arrhythmia (including QTC ≥ 440ms) and congestive heart failure above Grade 2 (New York Heart Association (NYHA) classification).
    3. Patients with active or uncontrolled severe infection (≥ CTC AE Level 2).
    4. Patients with a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
    5. Patients with poor control of diabetes (fasting blood glucose (FBG)>10mmol/L).
    6. Patients with urine protein ≥ ++ indicated by routine urine test, and confirmed 24-hour urine protein quantitation > 1.0 g.
    7. Patients with seizures requiring treatment.
12. Patients with bleeding tendency or medical history regardless of severity; Patients undergone bleeding events of a level ≥ CTCAE 3 within 4 weeks prior to the enrollment, and with unhealed wounds, ulcers or fractures.
13. Patients undergone venous thrombosis events currently or within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
14. Patients with a history of psychotropic drug abuse from which they are unable to abstain or with mental disorders.
15. Patients who have participated in other clinical trials of anti-tumor drugs within four weeks.
16. Patients with severe disease that threaten the safety of themselves or affect the completion of the study according to the investigators' judgment.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle
  the progression free survival of patients with extensive stage small cell lung cancer treated with anlotinib combined with EP/CE regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China